CLINICAL TRIAL: NCT01701791
Title: The Efficacy of Telemedicine for Improving Depression Outcomes in Primary Care
Brief Title: Telemedicine for Depression in Primary Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Responsible Party: Principal Investigator, Giovanni de Girolamo, M.D., Scientific Director, IRCCS Centro San Giovanni di Dio Fatebenefratelli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RF-2010-2316063
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Depression
Keywords: Depression; Primary care; Computerized decision support system; General practitioner
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Computerized Decision Support System (CDSS) (Experimental): GPs will use a CDSS with treatment algorithms, supervision from a consultant psychiatrist, and despatch to patients of reminders via mobile texting or automatic mobile (or landline) phone calls to improve adherence to the treatment prescribed.
  Interventions: Other: Computerized Decision Support System
- Treatment as usual (No Intervention): GPs will provide TAU, will make their own decisions and will therefore not use the CDSS. Patients will not receive any reminders.

INTERVENTIONS:
Other: Computerized Decision Support System
  Arms: Computerized Decision Support System (CDSS)

SUMMARY:
Background: In Italy, several recent studies found that a large percentage of patients attending Primary Care (PC) clinics meet criteria for at least one common mental disorder, as they show high rates of depression, anxiety, and co-morbid anxiety and depression. These patients may experience significant functional impairment and suffer from unexplained somatic symptoms, and often remain undetected and untreated. Consistent evidence for the effectiveness of organized care programs for depression, by improving quality of care and treatment adherence, is now available. Fundamental elements of these programs include algorithms to prompt the proper and timely implementation of evidence-based treatments, structured outcome assessment and systematic outreach. Telemedicine tools may represent a valuable strategy for improving depression outcomes in PC.

Aims: 1.To develop and employ computer-based assessment to more accurately and timely detect patient depression in PC settings; 2.To evaluate the feasibility and effectiveness of a care support program developed in conjunction with the PC-based assessment for patients suffering from depression, as based on two main objectives: 2a.To support GP decisions with treatment algorithms and improve the quality of GP and mental health service collaboration; 2b.To improve patient compliance and treatment adherence by using appropriate telecommunication tools and technologically advanced tools to conduct systematic routine assessment. Although much of this system will be computer-based, live telephonic and in-person contacts will also be included as needed.

Study Design: The study is a randomized controlled trial, involving four PC group clinics (GCs) located in two areas of Northern Italy. Two PC clinics will use the experimental protocol; the other two will serve as controls.

The study will compare two different conditions:

* Group 1 (experimental): GPs will use a Computer Decision Support System with treatment algorithms and advice and supervision from a consultant psychiatrist. Patients will receive reminders via mobile texting or automatic mobile (or landline) phone calls to improve adherence to the treatment prescribed.
* Group 2 (control): GPs will provide TAU, will make their own decisions and will therefore not use the CDSS. Patients will not receive any reminders. All enrolled patients will be administered and will fill in the IDS-SR at baseline, 3 and 6-months: the IDS-SR score will be used as a primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years
* PHQ-9 score of >or=14 at baseline
* IDS-SR score of >or=26 at baseline
* No filling of antidepressant medication prescription for 270 prior days
* Illiteracy or the lack of working telephone to receive reminders.

Exclusion Criteria:

* Current diagnosis of alcohol or substance dependence
* History of Bipolar Disorder determined by a baseline Composite International Diagnostic Interview (CIDI) screening scale of lifetime mania/hypomania
* Any current prescription for mood stabilizer or antipsychotic medication
* Female with positive pregnancy test
* General medical conditions which contraindicate antidepressant medications
* Clinical status requiring inpatient or day hospital treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-11; Primary Completion 2016-01 (Actual); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients reaching remission | 6 months
  The primary end-point will be the proportion of patients reaching remission by 6 months, as represented by an exit IDS-SR score of <or=12.

SECONDARY OUTCOMES:
Number of GP appointments actually attended during follow-up | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Balestrieri, M.D., Principal Investigator — IRCCS Centro San Giovanni di Dio Fatebenefratelli
Locations (4):
- Italy (4):
  - Health Telematic Network srl, Brescia, Brescia
  - IRCCS Centro San Giovanni di Dio Fatebenefratelli, Brescia, Brescia
  - Dipartimento di Scienze Mediche Sperimentali e Cliniche, Università di Udine, Udine, Udine
  - Marco B. Rocchi, Urbino

REFERENCES:
- [Derived] Balestrieri M, Sisti D, Rocchi M, Rucci P, Simon G, Araya R, de Girolamo G. Effectiveness of clinical decision support systems and telemedicine on outcomes of depression: a cluster randomized trial in general practice. Fam Pract. 2020 Nov 28;37(6):731-737. doi: 10.1093/fampra/cmaa077. PMID 32766705
- See also: Website of the Coordinating Centre — http://www.irccs-fatebenefratelli.it/